CLINICAL TRIAL: NCT05544474
Title: Definition of Surgical Technique of Lymphadenectomy and Complete Mesocolon Excision for Radical Right Colectomy: a Delphi Consensus
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Giuseppe Sigismondo Sica, Associate Professor, University of Rome Tor Vergata
Other Study IDs: 09/22
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert surgeon on radical right colectomy: Expert surgeon on radical right colectomy com pricing corresponding author/senior author from paper included in a preliminary systematic review on this topic Sica GS, Vinci D, Siragusa L, Sensi B, Guida AM, Bellato V, García-Granero Á, Pellino G. Definition and reporting of lymphadenectomy and complete mesocolic excision for radical right colectomy: a systematic review. Surg Endosc. 2022 Sep 12. doi: 10.1007/s00464-022-09548-5.
  Interventions: Other: Delphi questionnaire

INTERVENTIONS:
Other: Delphi questionnaire — An invitation email, including a link to the survey, will be sent to the panel of experts in the field of radical right colectomy. The Delphi questionnaire will be administered via www.surveymonkey.com.
  In the first survey, panel members will agree on surgical steps, definition of surgical steps and nomenclature for radical right colectomy In subsequent surveys, panel expert will agree on a common definition, nomenclature and reporting for right colectomy. Multiple rounds will be conducted until consensus is reached. After each round, the study team will calculate the agreement and distribution of responses. Likert responses will be dichotomized with positive values indicating agreement and neutral or negative values indicating disagreement.
  For the questions that do not reach a consensus of more than 70% in the first round or need further explanation, additional rounds of the survey may be performed.

SUMMARY:
A Delphi consensus to define surgical steps of lymphadenectomy and complete mesocolic excision for radical right colectomy

ELIGIBILITY:
Inclusion Criteria:

* Experts in the fields of radical right colectomy

Exclusion Criteria:

* Panelists who were not able to commit to all rounds of the modified Delphi process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Expert surgeon on radical right colectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-28 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Degree of consensus | 3 months
  The level of agreement for all statements achieving consensus from the expert panel; consensus is predefined as ≥ 80% of the panel rating a given statement

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome Tor Vergata, Rome, Italy

REFERENCES:
- See also: Sica GS, Vinci D, Siragusa L, et al. Definition and reporting of lymphadenectomy and complete mesocolic excision for radical right colectomy: a systematic review. Surg Endosc. 2022 Sep 12 — https://doi.org/10.1007/s00464-022-09548-5